CLINICAL TRIAL: NCT06603311
Title: Finite Treatment of Hepatitis Delta With Bulevirtide: Identification of Biomarkers Associated With Sustained Control of HDV Infection
Acronym: BUL-STOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: German Liver Foundation (DLS) (Unknown); HepNet Study House, German Liverfoundation (Network)
Responsible Party: Principal Investigator, Wedemeyer, Hans Heinrich Prof. Dr., Prof. Dr. Heiner Wedemeyer, Hannover Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BUL-STOP
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Compensated Liver Disease (Disorder); Hepatitis D, Chronic
Keywords: Bulevirtide; HDV; Biomarkers; compensated liver disease
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Intervention Model Description: After discontinuation of the standard treatment of patients with compensated liver disease and chronic hepatitis delta in subjects who received BLV for at least 48 weeks at the discretion of their treating physicians and have reached HDV RNA below 100 IU/ml for at least 24 weeks patients will followed-up for 48 weeks to identify the diagnostic value of biomarkers associated with HDV RNA relapse after stopping BLV and to evaluate the concept of finite BLV treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with compensated liver disease and HDV with prior Bulevirtide treatment (Experimental): Adults with compensated liver disease who have been treated for chronic HDV infection with bulevirtide (BLV) for at least 48 weeks and reached HDV RNA below 100 IU/ml for at least 24 weeks will finite their BLV treatment. Patients will be followed up for 48 weeks to identify promising biomarkers associated with HDV control after stopping BLV and to evaluate the safety of the novel concept of finite BLV treatment in this group of patients
  Interventions: Other: Stop Treatment with Bulevertide in patients with compensated liver disease and chronic HDV infection

INTERVENTIONS:
Other: Stop Treatment with Bulevertide in patients with compensated liver disease and chronic HDV infection — Stop Treatment with Bulevertide in patients with compensated liver disease and chronic HDV infection who have been treated for at least 48 weeks and reached HDV RNA below 100 IU/ml for at least 24 weeks.

SUMMARY:
Finding biomarkers for stopping bulevirtide treatment of patients with hepatitis delta

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm, discontinuation study in which patients who have been treated with BLV for at least 48 weeks, are intentionally discontinued from the treatment.

Currently, the treatment duration has not yet been defined and BLV can be given as long as a clinical benefit; is evident. In patients with advanced liver disease, maintenance treatment is recommended by most experts.

In pivotal phase II studies in which patients were treated with BLV for 24-48 weeks, some patients (10-20%) maintained a reduced HDV viral load with normal liver enzymes after the end of treatment (Wedemeyer et al., 2018, 2019, 2020). However, it is completely unclear which patients are able to control HDV infection without antiviral therapies. Biomarkers would be needed to identify patients in whom treatment can stopped safely. This is even more important because HDV flares can be life-threatening in the event of a relapse after stopping BLV. Thus, the main aim of this study is to explore biomarkers in blood and liver associated with maintained virological control after at least 24 weeks of HDV-RNA levels below 100 IU/ml, with at least 2 tests plus one test at screening, on BLV treatment. The investigators hypothesize that biomarker-based criteria should be able to identify patients with a sustained immune control. This information would be highly relevant to personalize treatment duration (or stopping) of BLV treatment, could reduce long-term disease burden, would enable safer treatments and also reduce treatment costs. Within the proposed systematic, unbiased study the investigators follow a broad screening for biomarkers that may be suitable to discriminate in a first step between patients that will experience a virological relapse (HDV RNA above 1000 IU/ml) after discontinuation of treatment and those without.

The investigators plan to include 20 patients in this study. These patients have to have received BLV treatment for at least 48 weeks and have to show HDV-RNA levels below 100 IU/ml in two repeated tests plus one test at screening, for at least 24 weeks while still being on treatment. Treatment will be stopped with the beginning of the study and patients will be followed for 48 weeks. It is expected that up to 14 patients will maintain HDV-RNA control (HDV-RNA below 1000 IU/ml). The other patients are expected to experience a virological relapse. Treating physicians should consider to re-initiate BLV at HDV-RNA levels of above 1000 IU/ml.

The aim of the study is to identify biomarkers that are associated with maintained virological response and could therefore be further investigated as predictive markers for treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Men, women, inter/diverse* aged ≥ 18 years
2. Signed written informed consent from subject
3. Chronic hepatitis delta
4. Stable and continued NUC treatment of the underlying HBV infection
5. Previous interferon treatment must have stopped at least 6 months before the start of BLV monotherapy
6. Previous immunosuppressant therapy must have stopped at least 6 months before the start of BLV therapy
7. BLV treatment for at least 48 weeks
8. HDV-RNA below 100 IU/ml under BLV treatment for at least 24 weeks. Patients should have had at least 2 tests with HDV-RNA below 100 IU/ml plus one test with HDV-RNA below 100 IU/ml+ at screening.
9. ALT level below 1.5 fold ULN

Exclusion Criteria:

1. Patients with decompensated liver cirrhosis (transient mild deviations in liver function parameters are acceptable at the discretion of the investigator) or history of decompensated liver cirrhosis (patients with minimal perihepatic ascites could be included at the discretion of the investigator)
2. Hepatocellular carcinoma (HCC)
3. Thrombocytopenia (platelet count below 90.000/µl)
4. Participation in another interventional clinical trial (other investigational drugs or devices at the time of enrolment or within 30 days prior to enrolment)
5. Any additional medical reason not to stop BLV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of biomarker on HDV-RNA relapse at week 48 | week 48
  All primary analysis will be carried out in the FAS. All patients will be categorized into two subgroups based on HDV-RNA relapse (yes/no) at week 48:
  1. HDV-RNA relapse: HDV-RNA ≥ 1000 IU/ml at any time point up to week 48
  2. No HDV-RNA relapse: HDV-RNA above 1000 IU/ml at all time points up to week 48 For the primary analysis, patients with missing HDV-RNA relapse outcome will be imputed with HDV-RNA relapse. Patients who re-initiated bulevirtide will be analysed as having a HDV-RNA relapse independent of their actual relapse status.

SECONDARY OUTCOMES:
Re-initiation of Bulevirtide (BLV) | week 48
  Number of patients who had to re-initiate treatment (all-cause)
Change in QoL | week 48
  Change in QoL between screening and end-of-study, as assessed by questionnaires
Alanine transaminase (ALT) values below 1.5x the upper limit of normal (ULN) at week 48 | week 48
  Number of patients with ALT values below 1.5 ULN at week 48 post treatment stop.
Alanine transaminase (ALT) values below 1.5x the upper limit of normal (ULN) at week 24 | week 24
  Number of patients with ALT values below 1.5 ULN at week 24 post treatment stop.
HDV-RNA below 100 IU/ml at week 48 | week 48
  Number of patients with HDV-RNA below 100 IU/ml at week 48 after the stop of BLV treatment
HDV-RNA below 100 IU/ml at week 24 | week 24
  Number of patients with HDV-RNA below 100 IU/ml at week 24 after the stop of BLV treatment

OTHER OUTCOMES:
Liver-related Events | week 48
  Development of liver-related events (decompensation, HCC, portal vein thrombosis)
Alanine transaminase (ALT) flares | week 48
  ALT flares after discontinuation of BLV, defined as ALT increases more than 5x upper limit of normal (ULN) at any time during the 48 weeks of follow-up after the discontinuation of BLV treatment.

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - University Hospital Heidelberg; Department of Internal Medicine IV: Gastroenterology, Hepatology, Infectious Diseases, Poisoning, Heidelberg, Baden-Wurttemberg
  - University Hospital Frankfurt; Medical Clinic 1, Frankfurt am Main, Hesse
  - Hannover Medical School; Department of Gastroenterology, Hepatology, Infectious Diseases and Endocrinology, Hanover, Lower Saxony
  - Charité - University Hospital Berlin (Campus Virchow-Clinic); Department of Hepatology and Gastroenterology, Berlin
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico; Division of Gastroenterology and Hepatology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No